CLINICAL TRIAL: NCT00370838
Title: Comparison of Keppra and Clonidine in the Treatment of Tics in Children With Tourette Syndrome
Brief Title: Comparison of Keppra and Clonidine in the Treatment of Tics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Harvey S. Singer (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor-Investigator, Harvey S. Singer, Haller Professor of Pediatric Neurology, Johns Hopkins University
Organization: Johns Hopkins University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TSkepclon
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Results first posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Tic Disorders; Tourette Syndrome
Keywords: Tics; Tourette syndrome; levetiracetam; clonidine
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome; Tics | interventions — Levetiracetam; Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levetiracetam (Experimental): Levetiracetam (Keppra) is used in one phase of this cross-over study.
  The initial dose of levetiracetam was 10 mg/kg/day, divided twice daily (rounded to the closest unit of 250 mg). The dose was increased weekly by 5-10 mg/kg/day, to a maximum dose of 50 mg/kg/day (or 2,500 mg/day), if deemed necessary for tic suppression. In any individual, dose escalation may have proceeded more slowly, or the dose may have been reduced as necessary. No changes in dosage occurred during the final week of either treatment phase.
  Interventions: Drug: Levetiracetam
- Clonidine (Active Comparator): Clonidine is used in one phase of this cross-over study.
  The initial dose of clonidine was 0.05 mg, twice daily. If needed for tic suppression, the dose was increased weekly by 0.05-0.1 mg, with a maximum dose of 0.4 mg per day. In any individual, dose escalation may have proceeded more slowly, or the dose may have been reduced as necessary. No changes in dosage occurred during the final week of either treatment phase.
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Levetiracetam — The initial dose of levetiracetam was 10 mg/kg/day, divided twice daily (rounded to the closest unit of 250 mg). The dose was increased weekly by 5-10 mg/kg/day, to a maximum dose of 50 mg/kg/day (or 2,500 mg/day), if deemed necessary for tic suppression. In any individual, dose escalation may have proceeded more slowly, or the dose may have been reduced as necessary. No changes in dosage occurred during the final week of either treatment phase.
  Other Names: Levetiracetam (Keppra)
  Arms: Levetiracetam
Drug: Clonidine — The initial dose of clonidine was 0.05 mg, twice daily. If needed for tic suppression, the dose was increased weekly by 0.05-0.1 mg, with a maximum dose of 0.4 mg per day. In any individual, dose escalation may have proceeded more slowly, or the dose may have been reduced as necessary. No changes in dosage occurred during the final week of either treatment phase.
  Other Names: Catapres
  Arms: Clonidine

SUMMARY:
The goal of this study is to confirm that levetiracetam has a better tic-suppressing profile than that of the widely used tic-suppressing medication, clonidine. More specifically, the investigators hypothesize that in a 15 week placebo run-in, double-blind, medication cross-over trial; levetiracetam will be more effective and have fewer side-effects than clonidine.

DETAILED DESCRIPTION:
This is a randomized, double-blind, 15 week (two treatment phase), 1 week run-in, cross-over study, in which the same patient receives 6 weeks of treatment with levetiracetam and a 6 week treatment course with clonidine, separated by a two week medication wash-out. The investigators plan to enroll twenty patients between the ages of 7 to 19 years with moderate to moderately-severe Tourette syndrome or chronic motor/vocal tics. The recruitment period is expected to be approximately 12 months (total study length of about 18 months). The study will begin with a screening evaluation to ensure that each subject satisfies all eligibility criteria, to allow subjects to become familiar with our assessment procedures, and to obtain informed consent. Following a baseline visit, there will be a one week "run-in" treatment period in order to screen for high placebo responders, in which all subjects will receive placebo. If the patient's tic severity score fails to improve he/she will begin the double blind treatment period (levetiracetam/clonidine), that will last for six weeks followed by a two week wash out period, and then by a second double blind treatment period (clonidine/levetiracetam) for an additional six weeks. A statistician not involved with the care of the subjects will be responsible for randomization. A six week trial treatment was chosen to allow for an adequate drug response period. Patients will be followed by phone at weekly intervals throughout the study and will be formally evaluated at the beginning and end of each treatment phase. At the completion of the study, patients/parents will be given the opportunity to continue a successful treatment.

The primary outcome measure is the Yale Global Tic Severity Scale (YGTSS): A semi-structured clinical interview designed to measure current tic severity. Other outcome measures will include the Clinical Global Impression-Improvement Scale (CGI-I), the Child Yale-Brown Obsessive-Compulsive Scale (CYBOCS), the DuPaul Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale, Child Depression Inventory (CDI), Multi-Dimensional Anxiety Scale for Children (MASC), and an expanded Pittsburgh Side-Effect Scale.

Subjects will be recruited from the Tourette Syndrome Clinic at the Johns Hopkins Hospital. This clinic, directed by Dr. Harvey Singer, currently follows more than 1000 chronic tic patients and averages 4 new referrals every week. The clinic staff has a longstanding successful record of designing and completing therapeutic protocols for the treatment of tics.

Inclusion Criteria: see below

Exclusion Criteria: see below

Procedures:

i) Screening visit: Determination of diagnostic eligibility criteria (medical history and complete physical examination; evaluation of tic severity, screening of females who have begun to menstruate with a urine pregnancy test, familiarization with assessment procedures, and obtaining informed consent. The urine pregnancy test will be obtained in females over 12 years of age. Parents will be told the results of these tests. If the patient is uncomfortable with our telling the results of the pregnancy test to her parent(s), then they may decide not to take part in this study.

ii) Baseline Visit (Day 0): Evaluation prior to the run-in (placebo) phase will include weight, heart rate, blood pressure, respiratory rate, rating scales for: tics, the Yale Global Tic Severity Scale (YGTSS) and Childhood Global Impression-TS (CGI-TS); adverse effects, the Pittsburgh Side-Effect Rating Scale; obsessive-compulsive problems, Child Yale-Brown Obsessive Compulsive Scale (CY-BOCS; attention deficit hyperactivity disorder, DuPaul ADHD Rating Scale, depression, Child Depression Inventory- Short Version (CDI-S); anxiety, the Multidimensional Anxiety Scale for Children (MASC; and episodic outbursts, Rage Attack Rating Scale.

iii) Run-in Placebo Phase (days 0-7): Immediately after the baseline visit, the subject is started on placebo treatment for a one week period. All subjects will receive 1 capsule twice a day; capsules will be similar in appearance to that used in the drug treatment phase. The Run-in phase has been added to eliminate subjects whose treatment outcome could be influenced by only a transient exacerbation of tics or by the exposure to non-pharmacologic treatment.

a) Post- Run in Period Evaluation (day 8): Subjects will return for a re-evaluation of symptoms, emphasis will be placed on rating scales for: tics, the Yale Global Tic Severity Scale (YGTSS) and Childhood Global Impression-TS (CGI-TS); and adverse effects, the Pittsburgh Side-Effect Rating Scale. If there is no tic improvement following the receipt of placebo, the patient will move on to the treatment phase of the study. In contrast, if tic symptoms are reduced by more than 15% or significant side effects are reported, all treatment will be discontinued and the subject will be withdrawn from the study.

iv) Treatment phases (days 8 50 and days 65 107): A computer generated unequal randomized scheme will be used to assign patients to either levetiracetam or clonidine in the initial treatment phase. Research Pharmacy at Johns Hopkins will be responsible for packaging levetiracetam (supplied by UCB) and clonidine (purchased), randomizing its allocation, and distributing the medication. Levetiracetam and clonidine will be repackaged in look-alike capsules with different dosage levels: levetiracetam, 250 milligrams (mg) or 500 mg and clonidine, 0.05 mg or 0.1 mg. Patients will receive a six week supply of medication at the first treatment phase visit (day 8) and at the beginning of the second treatment phase (day 63). A study physician (Dr. Harvey Singer) will be responsible for changing medication dosage and monitoring side-effects. A Safety Monitoring Board has been established to oversee medication use and monitor side-effects.

1. Levetiracetam: The starting dose of levetiracetam will be 10 mg/kg/day for one week; administered as 5 mg/kg twice a day (B.I.D.)(rounded to the closest unit of 250 mg). If needed for tic suppression, the dose will be increased weekly by 5-10 mg/killigrams(kg)/day. The maximum dose will be 50 mg/kg/day (administered as 25 mg/kg BID), with a maximum dose of 2,500 milligrams per day. For reference, doses from 10 to 60 mg/kg/day of levetiracetam are currently being used in pediatric studies for the treatment of seizures and up to 2000 mg in TS children with a mean age of 12 years. In any individual subject, dose escalation may proceed more slowly, or the dose may be reduced if necessary. No changes in dosage will be made during the final week of both treatment phases.
2. Clonidine: The starting dose of clonidine will be 0.05mg BID for one week. If needed for tic suppression, the dose will be increased weekly by 0.05-0.1 mg. The maximum dose will be 0.4 mg (administered as 0.2 mg BID).

iv) Wash out phase: Between the two treatment phases, medication will be tapered over a ten day period. Levetiracetam will be tapered at the end of each treatment phase by 5-10 mg/kg/day every third day. The half life of levetiracetam is approximately 7-8 hours in healthy volunteers, 5 8 hours in epileptic patients, and about 10 hours in the elderly. Clonidine will be tapered by 0.05 - 0.1 mg every third day. Subjects will be off medication for 5 days before starting the second phase of the cross over study.

v) End of study drug taper: At the completion of the second treatment phase, medication will be tapered over a ten-day period, reducing the medications in equal proportions every third day.

vi) Early stopping rules: Subjects may be withdrawn from the study at any time at the discretion of the subject, attending physician, or investigator.

1. The investigator decides the subject should be withdrawn. This decision could be made because of an adverse effect or a failure to comply with the study protocol.
2. The subject or his/her personal physician requests that the subject be withdrawn from the study.
3. The subject, for any reason, requires treatment with another therapeutic agent that could conflict with the use of levetiracetam or clonidine.
4. A Drug Safety Monitoring Board will monitor side effects and assist in determining whether a subject should be withdrawn from the trial. Members of this board are full time Johns Hopkins Hospital faculty members and epilepsy fellows with experience in the use of levetiracetam. The Board will have access to the randomization codes maintained by the statistician. A quarterly update meeting will be scheduled for the Monitoring Board with topics to be reviewed including the number of subjects, dosage schedules, side effects, and therapeutic responses. Significant adverse events will be reported to the sponsor Union chimique belge, Inc (UCB, Inc), Johns Hopkins Joint Committee on Clinical Investigation (JCCI), and Food and Drug Administration (FDA) within 24 hours.

vii) Evaluations: This is a 15 week study. Telephone evaluations will be performed by the blinded Research Assistant on day 14, 21, 28, 35, 42, 70, 77, 84, 91, and 98. At each telephone session clinical response, possible side effects, drug compliance, and medication adjustment will be discussed. Subjects will be formally evaluated at 4 separate times including baseline (day 0), at end of the run-in phase (day 8), end of the first treatment phase (day 49), at end of the drug wash out period (day 63), and at end of the study (day 105). Evaluations at each visit by the Research Assistant will include vital signs, weight, and an assessment of side effects using the Pittsburgh side effects scale. The blinded outcome evaluator, Dr. Harvey Singer, will administer and score the YGTSS, CGI I, DuPaul ADHD scale, CY BOCS, CDI S, and MASC. In addition, at each visit a pill count will be done to assure compliance.

C. Outcomes Measures:

i) Yale Global Tic Severity Scale (YGTSS): The YGTSS is a semi-structured clinical interview designed to measure current tic severity [Leckman et al., 1989]. This scale consists of the separate rating of severity for motor (total motor, 0 to 25) and vocal (total vocal, 0 to 25) tics. Ratings are made along 5 discriminant dimensions, on a scale of 0 to 5 for each including number, frequency, intensity, complexity, and interference. Summation of these scores (i.e., 0 to 50) provides a Total Tic Score (TTS) which will be the primary outcome measure. The YGTSS also contains a separate ranking of impairment (Tic Impairment Score or TIS), with a maximum of 50 points, based on the impact of the tic disorder on areas such as self esteem, family life, social acceptance, and school scores. Because the focus of this study is to evaluate the impact of levetiracetam and clonidine on tics and because the TIS may incorporate other components of TS, the Total Tic Score (TTS) has been selected as the primary outcome measure.

ii) Clinical Global Impression-Improvement (CGI-I): The CGI-I is used to compare current severity to baseline. A score of 1 corresponds to "very much improved; @ 2 equals "much improved;" 3 denotes minimal change; and 4 represents "no change." Scores above 4 are used to indicate deterioration, i.e., 5 equals "minimally worse;" 6 is "much worse;" and 7 is "very much worse."

iii) Child Yale-Brown Obsessive Compulsive Scale: The severity of OCD will be evaluated using the Child Yale-Brown Obsessive Compulsive Scale (CY-BOCS) [Scahill et al, 1997]. Obsessions and compulsions are rated on 5 separate scales yielding three summary scores: Obsessions (0-20), Compulsions (0-20) and a Total score (0-40). The CY-BOCS is the most widely used instrument to assess the severity of obsessive-compulsive symptoms in research studies involving children. It includes a checklist of specific obsessions and compulsions followed by examiner ratings of time spent, interference, distress, resistance and control over the obsessions and compulsions assessed independently. The CY-BOCS has well established psychometric properties.

iv) DuPaul ADHD Rating Scale: The presence of ADHD symptoms will be assessed using the DSM-IV version of the ADHD rating scale developed by DuPaul. This scale incorporates the symptom items for ADHD from the DSM into a rating scale format that quantifies symptom severity. Each item is rated as not at all, just a little, pretty much, and very much (0, 1, 2, and 3). This scale has been normed in large clinical and community samples and has excellent psychometric properties including a test-retest reliability over a 2-week period of 0.93 and significant correlations with direct observations of classroom behavior.

v) Child Depression Inventory-Short Version (CDI-S): Depression severity will be rated by using the Child Depression Inventory-Short Version (CDI-S. This 10 item scale takes about 5 minutes to complete. It has excellent psychometric properties and is designed for repeated administrations over time.

vi) Multidimensional Anxiety Scale for Children (MASC): The child's anxiety will be followed using the multidimensional Anxiety Scale for Children (MASC) and is now considered the preferred instrument for rating childhood anxiety.

vii) Adverse effects: Side effects will be assessed by an expanded Pittsburgh Side Effect Scale modified to include side effects of levetiracetam and clonidine. Significant adverse events will be reported to the UCB, JCCI, and FDA within 24 hours.

D. Open Label Continuation:

At the completion of the study the subject will be given the option of continuing either levetiracetam or clonidine in an open labeled fashion. This will be enabled by having the subject seen by another physician who will have access to the study codes. This physician will continue to follow the subject until the entire study is completed. For members of the research team, the treatment code will not be broken until all subjects have completed the protocol.

IV. Analytical Strategies A. Inclusion of a Run-in phase: The Run-in phase has been added to eliminate subjects whose treatment outcome could be influenced by a transient exacerbation of tics or by the exposure to non-pharmacologic treatment.

B. Power calculations: As described, this is a pilot randomized, double-blind, placebo-controlled, cross-over project in which the investigators plan to enroll twenty patients between the ages of 7-19 years with Tourette Syndrome. Subjects with moderate to severe TS will be enrolled in this treatment protocol. Data from randomized, double-blind, placebo-controller trials of tics suggest that 6.0 points in the YGTSS total tic score is a reasonable estimate of the standard deviation of this outcome variable in the population of interest. The investigators estimate that approximately 19 subjects will provide a desired power of 0.9 to detect a difference of 4.2 points in the mean 6-week change in YGTSS total tic score between the two treatment arms, using a two-tailed t-test and a 5% level of significance.

C. Statistical evaluations: The primary outcome measure is effective tic suppression as determined by the difference in Total Tic scores between treatment arms for levetiracetam and clonidine. Secondary outcome measures include the Tic Impairment Score, the Total YGTSS score, and the CGI-I. Data will be compared both as a change in absolute test score and as a percentage from baseline. Unpaired Student's t-tests will be used to compare treatment and placebo groups across all clinical variables at baseline. A paired t-test with a 95% confidence interval will be used to compare changes in outcome measures from baseline to endpoint between the two treatment groups (levetiracetam and clonidine) regardless of treatment order. Using a secondary assessment (Analysis of Variance (ANOVA) with levels within respective classes containing subjects completing study, 2 treatments, and 2 periods), the investigators will analyze each outcome measure as a two-period (days 8 to 49 or 63 to 105), two-treatment, two-sequence design with a test for the effects of treatment, first or second period, and treatment by period interaction. To evaluate the effect of levetiracetam and clonidine on blood pressure, pulse, weight, DuPaul ADHD scale, CYBOCS, CDI-S, and MASC, the investigators will conduct a series of repeated measures ANOVA to examine differences in each group across time. Statistical significance for all analyses will be set at alpha=0.05 for a two-tailed test. This protocol format has been used effectively in a prior study of baclofen and levetiracetam.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in this study if they meet the following criteria:

* Tourette syndrome criteria based on the TS Classification Study Group [1993], which includes onset before 18 years, multiple involuntary motor tics, one or more vocal tics, a waxing and waning course, the gradual replacement of old symptoms with new ones, the presence of tics for more than one year, the absence of other medical explanations for tics, and observation of tics by a reliable examiner;
* Age 7 to 19 years, either gender;
* Observable tics, achieving a minimum score of > 22 on the Total Tic score of Yale Global Tic Severity Scale (YGTSS);
* Tic symptoms severe enough to warrant therapy;
* The concurrent use of other tic-suppressing medications will be permitted, if the subject has been on a stable dose for more than three weeks and agrees to maintain a constant dosage throughout the study;
* Tics are not controlled with current medication or individuals are tic suppressing drug naive.

Exclusion Criteria:

Exclusion criteria include the following:

* Secondary tics;
* Significant medical illness
* Current major depression, generalized anxiety disorder, separation anxiety disorder, psychotic symptoms (based on clinical evaluation), pervasive developmental disorder, autism, mental retardation (I.Q. less than 70), anorexia/bulimia, or substance abuse. Subjects with co-morbid ADHD, obsessive compulsive disorder (OCD), and conduct disorder will not be excluded;
* pregnancy;
* Hypersensitivity to levetiracetam or clonidine;
* baseline weight of less than 25 kilograms.

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2007-02; Primary Completion 2008-07 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harvey S Singer, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 participants signed informed consent, but 2 participants were never randomized to treatment arm.
Groups:
- First Levetiracetam Then Clonidine: Participants first received levetiracetam: starting dose of 10 milligram/killigram/day, increased weekly by 5-10 milligram/killigram/day, to a maximum of 50 milligram/killigram/day (25 milligram/killigram twice a day; 2,500 mg per day).
  In the second period, participants received clonidine (days 65-107), packaged in look-alike capsules: starting dose was 0.05 milligrams twice a day, if needed, the dose increased weekly by 0.05-0.1 milligrams. The maximum dose was 0.4 milligrams (0.2 milligrams twice a day).
  Wash out phase: Between the two treatment phases, medication tapered over a ten day period: levetiracetam by 5-10 mg/kg/day every third day; clonidine by 0.05 - 0.1 mg every third day. Subjects were off medication for 5 days before starting the second phase of the cross over study.
  Taper: After the two treatment phases, medication tapered over a ten day period as in Wash-out phase (see above).
- Clonidine First, Then Levetiracetam: Participants first received clonidine, packaged in look-alike capsules: starting dose was 0.05 milligram (mg) twice a day, if needed, the dose increased weekly by 0.05-0.1 mg. The maximum dose was 0.4 mg (0.2 mg twice a day (BID)).
  In the second period, participants received levetiracetam: starting dose of 10 mg/killigram(kg)/day, increased weekly by 5-10 mg/kg/day, to a maximum of 50 mg/kg/day (25 mg/kg BID; 2,500 mg per day).
  Wash out phase: Between the two treatment phases, medication tapered over a ten day period: levetiracetam by 5-10 mg/kg/day every third day; clonidine by 0.05 - 0.1 mg every third day. Subjects were off medication for 5 days before starting the second phase of the cross over study.
  Taper: After the two treatment phases, medication tapered over a ten day period as in Wash-out phase (see above).
Period: Period 1 (Days 8-50)
Arm/Group | First Levetiracetam Then Clonidine | Clonidine First, Then Levetiracetam
Started | 7 | 3
Completed | 7 | 3
Not Completed | 0 | 0
Period: Washout (Days 51-64)
Arm/Group | First Levetiracetam Then Clonidine | Clonidine First, Then Levetiracetam
Started | 7 | 3
Completed | 7 | 3
Not Completed | 0 | 0
Period: Period 2 (Days 65-107)
Arm/Group | First Levetiracetam Then Clonidine | Clonidine First, Then Levetiracetam
Started | 7 | 3
Completed | 7 | 3
Not Completed | 0 | 0
Period: Taper
Arm/Group | First Levetiracetam Then Clonidine | Clonidine First, Then Levetiracetam
Started | 7 | 3
Completed | 7 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Levetiracetam First, Then Clonidine: Participants first received levetiracetam: starting dose of 10 milligram/killigram/day, increased weekly by 5-10 milligram/killigram/day, to a maximum of 50 milligram/killigram/day (25 milligram/killigram twice a day; 2,500 mg per day).
  In the second period, participants received clonidine (days 65-107), packaged in look-alike capsules: starting dose was 0.05 milligrams twice a day, if needed, the dose increased weekly by 0.05-0.1 milligrams. The maximum dose was 0.4 milligrams (0.2 milligrams twice a day).
  Wash out phase: Between the two treatment phases, medication tapered over a ten day period: levetiracetam by 5-10 mg/kg/day every third day; clonidine by 0.05 - 0.1 mg every third day. Subjects were off medication for 5 days before starting the second phase of the cross over study.
  Taper: After the two treatment phases, medication tapered over a ten day period as in Wash-out phase (see above).
- Total: Total of all reporting groups
Arm/Group | Levetiracetam First, Then Clonidine | Clonidine First, Then Levetiracetam | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 2 | 8
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 14.5 (6.4) | 16.0 (4.4) | 14.9 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 6 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Yale Global Tic Severity Scale (YGTSS):
Description: The YGTSS is a semi-structured clinical interview designed to measure current tic severity [Leckman et al., 1989], and consists of separate rating of motor (0-25) and vocal (0-25) tics. Ratings are made along 5 discriminant dimensions, scaled 0-5 for each including number, frequency, intensity, complexity, and interference. Total of these scores (0-50) is a Total Tic Score (TTS). The YGTSS contains an impairment ranking, 0-50 points, based on the impact of the tic disorder on areas such as self esteem, family life, social acceptance, and school. 0=no tics present; 100=most severe tics.
Time Frame: Baseline (Day 8 or Day 64), Final (6 weeks later: Day 50 or Day 106)
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Levetiracetam: Participants received levetiracetam in either first or second period of this study. The initial dose of levetiracetam was 10 mg/kg/day, divided twice daily (rounded to the closest unit of 250 mg). The dose was increased weekly by 5-10 mg/kg/day, to a maximum dose of 50 mg/kg/day (or 2,500 mg/day), if deemed necessary for tic suppression. In any individual, dose escalation may have proceeded more slowly, or the dose may have been reduced as necessary. No changes in dosage occurred during the final week of either treatment phase.
- Clonidine: Participants received clonidine in either the first or second phase of the study. The initial dose of clonidine was 0.05 mg, twice daily. If needed for tic suppression, the dose was increased weekly by 0.05-0.1 mg, with a maximum dose of 0.4 mg per day. In any individual, dose escalation may have proceeded more slowly, or the dose may have been reduced as necessary. No changes in dosage occurred during the final week of either treatment phase.
Arm/Group | Levetiracetam | Clonidine
Number analyzed (Participants) | 10 | 10
scores on a scale
  Baseline | 45.2 (12.7) | 48.7 (9.6)
  Final | 48.8 (21.8) | 43.1 (11.2)

2. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I):
Description: Clinical Global Impression-Improvement (CGI-I): The CGI-I is used to compare current severity to baseline. A score of 1 corresponds to "very much improved; 2 equals "much improved;" 3 denotes minimal change; and 4 represents "no change." Scores above 4 are used to indicate deterioration, i.e., 5 equals "minimally worse;" 6 is "much worse;" and 7 is "very much worse."
Time Frame: Baseline (Day 8 or Day 64), Final (6 weeks later: Day 50 or Day 106)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Levetiracetam | Clonidine
Number analyzed (Participants) | 10 | 10
scores on a scale
  Baseline | 4.1 (0.74) | 4.1 (0.6)
  Final | 4.1 (0.74) | 4 (0.5)

3. Secondary Outcome: Child Yale-Brown Obsessive Compulsive Scale (CY-BOCS):
Description: The severity of obsessive-compulsive disorder (OCD) is evaluated using the CY-BOCS [Scahill et al 1997]. Obsessions and compulsions are rated on 5 separate scales yielding three summary scores: Obsessions (0-20), Compulsions (0-20) and Total score (0-40). The CY-BOCS is the most widely used instrument to assess the severity of OCD symptoms in research studies. It includes checklist of specific obsessions and compulsions followed by examiner ratings of time spent, interference, distress, resistance and control over the obsessions and compulsions.0=no obsessions or compulsions; 40=most severe OC
Time Frame: Baseline (Day 8 or Day 64), Final (6 weeks later: Day 50 or Day 106)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Levetiracetam | Clonidine
Number analyzed (Participants) | 10 | 10
scores on a scale
  Baseline | 4.7 (5) | 3.1 (4.1)
  Final | 2.2 (3.7) | 3.2 (4.5)

4. Secondary Outcome: DuPaul Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale:
Description: The presence of Attention Deficit Hyperactivity Disorder (ADHD) symptoms are assessed using the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) version of the DuPaul ADHD rating scale, which incorporates the symptom items for ADHD from the DSM into a rating scale format that quantifies symptom severity. Each item is rated as not at all, just a little, pretty much, and very much (0, 1, 2, and 3). There are 18 items in total are summed, with a minimum score of 0 (meaning no inattention or hyperactivity) with a maximum score of 54 (severe inattention and hyperactivity).
Time Frame: Baseline (Day 8 or Day 64), Final (6 weeks later: Day 50 or Day 106)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Levetiracetam | Clonidine
Number analyzed (Participants) | 10 | 10
scores on a scale
  Baseline | 12.5 (10.3) | 12.6 (11.1)
  Final | 12.7 (10.6) | 11.9 (10.6)

5. Secondary Outcome: Multidimensional Anxiety Scale for Children (MASC):
Description: The child's anxiety will be followed using the multidimensional Anxiety Scale for Children (MASC) (Stallings and March, 1995) and is now considered the preferred instrument for rating childhood anxiety. It is a 39-item questionnaire, ranking each item as "Never", "Rarely", "Sometimes", or "Often" (0, 1, 2, 3). The sum of all responses yeilds a score (maximum MASC score is 117). A score of 0 represents no anxiety, and a score of 117 represents severe anxiety.
Time Frame: Baseline (Day 8 or Day 64), Final (6 weeks later: Day 50 or Day 106)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Levetiracetam | Clonidine
Number analyzed (Participants) | 10 | 10
scores on a scale
  Baseline | 32.9 (15.4) | 25.2 (17.1)
  Final | 27.5 (16.2) | 25 (14.7)

6. Secondary Outcome: Modified Pittsburgh Side Effect Scale
Description: Side effects will be assessed by an expanded (modified) Pittsburgh Side Effect Scale modified to include side effects of levetiracetam and clonidine. Significant adverse events will be reported to the UCB, JCCI, and FDA within 24 hours. Positive responses are tallied as "number of side effects" for the responding period.
Time Frame: Baseline (Day 8 or Day 64), Final (6 weeks later: Day 50 or Day 106)
Measure: Mean (Standard Deviation); unit: Number of Side Effects
Arm/Group | Levetiracetam | Clonidine
Number analyzed (Participants) | 10 | 10
Number of Side Effects | 2.1 (2.1) | 3.4 (4.5)

7. Primary Outcome: Total Tic Score
Description: The TTS is a portion of the YGTSS [Leckman et al., 1989], and consists of separate rating of motor (0-25) and vocal (0-25) tics. Ratings are made along 5 discriminant dimensions, scaled 0-5 for each including number, frequency, intensity, complexity, and interference. Total of these scores (0-50) is a Total Tic Score (TTS). A score of 0 represent no tics present, a score of 50 represents the most severe tics in each category listed.
Time Frame: Baseline (Day 8 or Day 64), Final (6 weeks later: Day 50 or Day 106)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Levetiracetam | Clonidine
Number analyzed (Participants) | 10 | 10
scores on a scale
  Baseline | 22.7 (5.7) | 25.2 (4.3)
  Final | 23.6 (10.6) | 21.8 (4.4)

ADVERSE EVENTS:
Arm/Group | Levetiracetam | Clonidine
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=10) | Clonidine (N=10)
Irritability (General disorders) | 3 (7) | 2 (2)
Sad/depressed (General disorders) | 2 (4) | 1 (1)
Hyperactive (General disorders) | 2 (2) | 0 (0)
Tired/sleepy (General disorders) | 2 (2) | 5 (17)
Anxious (General disorders) | 3 (3) | 4 (4)
Lethargic (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (2) | 3 (3)
Dizzy (General disorders) | 1 (1) | 1 (2)
Aggression (Psychiatric disorders) | 2 (5) | 3 (3)
Stomache ache (General disorders) | 0 (0) | 2 (2)
Dry mouth (General disorders) | 1 (1) | 1 (1)
Insomnia (General disorders) | 2 (2) | 2 (5)
Loss of appetite (General disorders) | 1 (1) | 0 (0)
Sleepwalking (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No